CLINICAL TRIAL: NCT02772445
Title: Stroke Caregiver Empowerment
Acronym: STROKE-CARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Juleen Rodakowski, Assistant Professor, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PRO16020650
Record Dates: First submitted 2016-03-31; First posted 2016-05-13 (Estimated); Last update posted 2021-07-06 (Actual); Status verified 2021-07

CONDITIONS: Stroke
Keywords: Empowerment; Caregiver
MeSH Terms: conditions — Stroke; Empowerment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- STROKE-CARE Intervention (Experimental): In STROKE-CARE, caregivers will learn a problem-solving strategy. Participants will receive approximately 10 sessions by an occupational therapist in the home over a 5 week process.
  Interventions: Behavioral: STROKE-CARE

INTERVENTIONS:
Behavioral: STROKE-CARE — In STROKE-CARE, caregivers will learn a problem-solving strategy. They will (1) identify barriers to performance, (2) generate strategies to address barriers, and (3) apply these strategies to support care-recipients in occupations.

SUMMARY:
The purpose of this study is to refine STROKE-CARE for caregivers and explore changes in caregiver and care-recipient outcomes

DETAILED DESCRIPTION:
Individuals with disabilities rely heavily on unpaid family caregivers to help perform necessary occupations. The emotional and physical demands of caregiving often contribute to caregivers experiencing burden. Caregivers with burden are at-risk for poor health and a heightened risk of mortality. This is likely, in turn, to negatively impact care-recipient quality of life. The proposed study refines a behavioral intervention that teaches caregivers to facilitate problem solving over the course of daily activities. The long-term goal for this project is to establish an effective rehabilitation intervention that promotes caregiver health and well-being, which ultimately influences care-recipient health. This study will use an open-case series and a single-arm clinical trial to refine the intervention and examine caregiver and care-recipient response to the intervention. This research applies to the priorities and objectives of this research initiative through examination of a caregiver-centered, standardized intervention that is based on occupational theories and principles, investigating outcomes experienced by caregivers of individuals with cognitive deficits after stroke. Data from this pilot project will be used to design and obtain federal funding for a randomized controlled trial to examine the efficacy of the refined intervention on caregiver and care-recipient health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Primary caregiver for an individual post-stroke
* Live with the care-recipient
* Provide 1 hour of caregiving per day
* Subjective caregiver burden

Exclusion Criteria:

* non-English speaking
* Active treatment (chemotherapy, radiation therapy) for cancer
* Imminent placement of care-recipient into a nursing home or with another caregiver (within 6 months)
* Involvement in another clinical trial for caregivers

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-04; Primary Completion 2018-03 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
The proportion of caregivers that use the universal strategy in daily activities | after study completion, an average of 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No